CLINICAL TRIAL: NCT06700759
Title: Yoğun Bakım Ünitesinde Takip Edilen Hastalarda Gastrik Boşalmanın Abdominal Ultrasonografi Ile Değerlendirilmesi
Brief Title: Ultrasound Vs. Free Drainage for Gastric Volume in ICU Patients on Enteral Nutrition
Status: Completed | Type: Observational
Sponsor: Ilkay Ceylan (Other Government)
Responsible Party: Sponsor-Investigator, Ilkay Ceylan, MD, Bursa Yuksek Ihtisas Training and Research Hospital
Organization: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Other Study IDs: 2011-KAEK-25 2022/01-19
Record Dates: First submitted 2024-11-13; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Gastric Residual Volume
Keywords: ultrasonography; gastric residual volume; enteral feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Patients who received 18 hours of infusion feeding, 6 hours of waiting and one hour of drainage
- Group 2: Patients who received 5 hours of infusion feeding, 1 hour of waiting and one hour of drainage
- Group 3: Patients who were fed with continuous infusion for 24 hours and drained for one hour

SUMMARY:
This study aims to evaluate the compatibility of gastric volume (GV) measurements obtained through ultrasound with the free drainage method in intensive care patients receiving enteral nutrition under three different protocols. The study seeks to determine the consistency of GV measurements across these protocols to improve patient management in critical care settings.

DETAILED DESCRIPTION:
Adult patients hospitalized in intensive care unit due to cerebrovascular disease and receiving mechanical ventilator treatment were included in the study. Patients who were started on semi-solid nutritional solution (standard nutritional products of 1kcal/1 ml according to the comorbidities of the patients) via nasogastric (NG) 14 F polyurethane (PU) feeding catheter (BAXEN Medical, Spain) and reached the full calorie goal for at least 24 hours were included. Full dose calorie calculation of the patients was performed using the Harris-Benedict method (for women: 655.1+(9.56xweight (kg)) -(1.85xheight (cm)) -(4.68xage) for men: 66.5+(13.75xweight (kg)) +(5.03xheight (cm)) -(6.75xage). Feeding tube placement was confirmed with an AP radiograph taken before inclusion in the study.

Patients with shock due to any cause, abdominal surgery, GI bleeding, obstruction, suspected perforation, malabsorption syndrome, prokinetic use or diarrhea, patients with a BMI >35 according to last known height and weight, and pregnant patients (due to inability to achieve right lateral position) were excluded. In addition, patients who could not be imaged, whose feeding protocol was changed and whose vasopressor doses were increased were excluded from the study.

The amount of EN products administered to the patients, age, gender, body weight, height, body mass index (BMI), comorbidities, vasopressor therapy and dose administered during imaging were recorded.

ICU units have a physician-driven nutrition strategy, aiming for an adequate caloric and protein intake. Patients were divided into 3 groups according to implemented nutrition protocols. Ultrasonographic measurements were performed in 24-hour periods after the volume required for the target calorie intake.

Group 1: Patients who received 18 hours of infusion feeding, 6 hours of waiting and one hour of drainage Group 2: Patients who received 5 hours of infusion feeding, 1 hour of waiting and one hour of drainage Group 3: Patients who were fed with continuous infusion for 24 hours and drained for one hour Measurement of gastric volume

1. Measurement by GUSG Using the GE LOQIC P6 (GE healthcare, USA) ultrasound device available in clinic and a convex probe (2-5 MHz), the patient was placed in the right lateral position. To visualize the antrum, the probe was scanned in the sagittal plane in the epigastrium, sliding from left to right along the subcostal margins. The gastric antrum, aorta, superior mesenteric artery and inferior vena cava were visualized just below the left lobe of the liver with the pancreas posterior to it. For the calculation of cross-sectional antral area (CSA), the anterior-posterior diameter and cephalo-caudal diameter (measured 3 times and averaged) were measured from serosa to serosa by capturing the best image during peristaltic movements at the level of the aorta or inferior vena cava. The antral area was calculated according to the formula CSA=(AP×CC×π)/4 (π=3.14) developed by Bolondi et al.

   Two different formulas were then used to calculate GV by CSA. The first formula was proposed by Perlas et al.: Gastric volume (ml)=27+(14.6×right-lateral CSA)-1.28×age1. The second formula was developed by Tacken et al.: Gastric volume (ml)= 79.38+13.32 x right-lat CSA.
2. Measurement by drainage After gastric volume was evaluated by USG, the patient was placed in supine position, NG was connected to a drainage bag and gravity/free drainage was performed in all groups for one hour and the GRV values were recorded.

ELIGIBILITY:
Inclusion Criteria:

Age Range: Adult patients aged 18 years and older.

ICU Admission: The study will include only patients who are currently admitted to the Intensive Care Unit (ICU) due to cerebrovascular diseases

Receiving Enteral Nutrition: Patients must be receiving enteral nutrition through one of the three specified protocols.

Eligibility for Gastric Volume (GV) Measurement: Patients must be medically eligible for GV measurement via ultrasound.

Informed Consent: The patient or their legal representative must provide informed consent to participate in the study.

Exclusion Criteria:

Age Below 18: Patients under 18 years of age.

Pregnancy: Pregnant patients will be excluded due to potential risks or confounding factors related to pregnancy.

Gastrointestinal Surgery History: Patients with a recent history of gastrointestinal surgery, which may affect GV measurements, will be excluded.

Contraindications for Ultrasound: Patients with conditions that prevent safe or accurate ultrasound measurement (e.g., severe abdominal wounds or high abdominal obesity) will be excluded.

Inability to Tolerate Enteral Nutrition: Patients who are unable to receive enteral nutrition for any reason (e.g., severe intolerance, contraindications) will be excluded.

Lack of Informed Consent: Patients or their legal representatives who do not provide informed consent.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neurocritical care patients
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Agreement Between Ultrasound and Free Drainage for Gastric Volume Measurements | Gastric volume measurements will be conducted at 24 hours after initiating each enteral nutrition protocol
  Gastric volume will be measured in ICU patients using ultrasound imaging and the free drainage method. Agreement between the two methods will be evaluated using Bland-Altman analysis and Intraclass Correlation Coefficients (ICCs). The data will be reported as mean ± standard deviation for continuous variables and proportions for categorical data. Results will be aggregated across the three enteral nutrition protocols.

OTHER OUTCOMES:
complications | Complications will be recorded at 24-hour intervals during the ICU stay, up to a maximum of 7 days.
  Nutritional Complications: Evaluation of potential complications (e.g., aspiration, abdominal distantion etc.) associated with the protocols in light of GV measurements.

CONTACTS AND LOCATIONS:
Overall Officials: İlkay Ceylan, Principal Investigator — Bursa Yüksek İhtisas Training Hospital
Locations (1):
- Bursa Yüksek İhtisas Education and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data collected throughout the trial.
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Who Will Be Able to Access the Data:
  Access to the study data will be limited to authorized researchers affiliated with accredited academic or healthcare institutions who have a valid research purpose aligned with the study objectives.
  Regulatory authorities may also be granted access if required for compliance or validation purposes.
  What They Will Be Able to Access:
  De-identified individual participant data (IPD), including demographic data, primary and secondary outcome measures, and other relevant clinical data collected during the study.
  Supporting documentation, such as the study protocol, statistical analysis plan, and informed consent forms.
  How They Will Be Able to Access It:
  Data will be provided through a secure data-sharing platform or repository, with access granted upon approval by the study's data access committee.
  Interested researchers must submit a data access request that includes an agreement to maintain data confidentiality